CLINICAL TRIAL: NCT04356092
Title: Feasibility of 2D Perfusion DSA With Custom-made, Color-coded Software for the Quantification of Foot Perfusion Following Infrapopliteal Angioplasty
Brief Title: 2D Perfusion DSA for the Quantification of Infrapopliteal Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Assistant Professor in Interventional Radiology, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 264/12.04.2017
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Ischemia Limb
Keywords: Infrapopliteal angioplasty; Tissue perfusion; Quantification

STUDY DESIGN:
Intervention Model Description: In total, 7 consecutive patients were included in the study. The 2D-perfusion imaging and analysis of the DICOM files were performed after revascularization.
Masking Description: 2D-perfusion imaging and analysis of the DICOM files was performed after revascularization, by an investigator blinded to the name of the patient or the result of the angioplasty procedure. The participant was also blinded to the results of the perfusion outcomes during follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perfusion (Experimental): Consecutive patients scheduled to undergo infrapopliteal angioplasty or stenting, or both, as part of their standard treatment for Rutherford-Becker class 5 and 6 chronic limb-threatening ischemia, were included in the study. All procedures were performed using local anesthesia. An antegrade access was used in all patients followed by the deployment of a 5 or 6 Fr arterial sheaths. A semi-lateral foot projection was preferred and the pre-revascularization DSA of the foot was performed via a 5 Fr angiographic catheter placed at the distal third of the popliteal artery. Following revascularization of one or more tibial arteries, the catheter was placed at the same popliteal segment and post-procedural DSA of the foot was performed following the exact pre-revascularization injection protocol at the same semi-lateral projection. The 2D-perfusion imaging and analysis of the DICOM files was performed after revascularization.
  Interventions: Diagnostic Test: 2D perfusion digital subtraction angiography of the foot.

INTERVENTIONS:
Diagnostic Test: 2D perfusion digital subtraction angiography of the foot. — 2D perfusion digital subtraction angiography of the foot was performed after infrapopliteal angioplasty and Perfusion Blood Volume (PBV), Mean Transit Time (MTT), and Perfusion Blood Flow (PBF) maps were extracted by analyzing Time-Intensity Curves and signal intensity on the perfused vessel mask.
  Other Names: Infrapopliteal angioplasty

SUMMARY:
A custom-made, 2D-perfusion digital subtraction angiography (PDSA) algorithm has been designed and implemented towards foot perfusion quantification following endovascular treatment of critical limb ischemia (CLI), in order to assist intra-procedural decision-making and enhance clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective, single-center, study investigating the feasibility of 2D-PDSA using newly-developed, non-commercially available, color-coded software for the quantification of foot perfusion following infrapopliteal angioplasty for the treatment of CLI. In total, 7 consecutive patients scheduled to undergo infrapopliteal endovascular treatment of CLI were enrolled. Perfusion Blood Volume (PBV), Mean Transit Time (MTT), and Perfusion Blood Flow (PBF) maps were extracted by analyzing Time-Intensity Curves and signal intensity on the perfused vessel mask. Mean values calculated from user-specified ROIs on perfusion maps were employed to evaluate the patient's pre- and post- endovascular treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescheduled for infrapopliteal angioplasty due to chronic limb-threatening ischemia.
* Written informed consent obtained

Exclusion Criteria:

* Image post-processing not feasible due to significant motion artifacts produced during DSA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-07-14 (Actual)

PRIMARY OUTCOMES:
Change in Perfusion Blood Volume (PBV) | Ten minutes before and five minutes after the intervention
  PBV calculated on subtraction images and pre- and post-procedural values were compared using the proposed 2D perfusion DSA software.
Change in Mean Transit Time (MTT) | Ten minutes before and five minutes after the intervention
  MTT calculated on subtraction images and pre- and post-procedural values were compared using the proposed 2D perfusion DSA software.
Change in Perfusion Blood Flow (PBF) | Ten minutes before and five minutes after the intervention
  PBF calculated on subtraction images and pre- and post-procedural values compared using the proposed 2D perfusion DSA software.

SECONDARY OUTCOMES:
Major amputation rate | Six months
  The rate of above the knee target limb amputation
Procedure-related complications | 30 days
  Complications noted during and after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Karnamatidis, MD, PhD, Study Chair — Patras University Hospital, Rion, Greece; George Kagadis, PhD, FAAPM, Principal Investigator — University of Patras, Greece
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Kagadis GC, Tsantis S, Gatos I, Spiliopoulos S, Katsanos K, Karnabatidis D. 2D perfusion DSA with an open-source, semi-automated, color-coded software for the quantification of foot perfusion following infrapopliteal angioplasty: a feasibility study. Eur Radiol Exp. 2020 Sep 2;4(1):47. doi: 10.1186/s41747-020-00176-z. PMID 32875390